CLINICAL TRIAL: NCT02468843
Title: Novel Stimulation Patterns and Personalized Deep Brain Stimulation for the Treatment of Dystonia
Brief Title: Novel Stimulation Patterns for the Treatment of Dystonia
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB201500366
Record Dates: First submitted 2015-06-03; First posted 2015-06-11 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Dystonia; Cervical Dystonia
Keywords: Deep brain stimulation; DBS; Dystonia; DYT1
MeSH Terms: conditions — Dystonia; Torticollis; Dystonia musculorum deformans type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Biphasic DBS stimulations: Subjects in this group with have Biphasic DBS stimulation setting performed, Unified Dystonia Rating Scale (UDRS), and Burke-Fahn- Marsden scale (BFMDRS), tremor accelerometer, kinesia accelerometer, and GaitRite walking assessments performed.
  Interventions: Device: Biphasic DBS stimulation; Other: Unified Dystonia Rating Scale; Other: Burke-Fahn- Marsden scale

INTERVENTIONS:
Device: Biphasic DBS stimulation — The following protocol will be followed for each subject. In between, baseline and novel stimulation settings there will be a 30-minute washout period with DBS in the off state.
  1. Current best/optimized DBS setting (considered "baseline")
  2. DBS off for 30 minutes
  3. Biphasic pulse stimulation mode (immediate assessment)
  4. Biphasic pulse stimulation mode (assessment at 1h)
  5. Biphasic pulse stimulation mode (assessment at 2h)
Other: Unified Dystonia Rating Scale — Neurologist use the UDRS to determine the severity and duration of dystonia on 14 body areas.
  Other Names: UDRS
Other: Burke-Fahn- Marsden scale — Neurologist use the BFMDRS to rate the severity of dystonia in 9 regions of the body.
  Other Names: BFMDRS

SUMMARY:
Deep brain stimulation (DBS) is an effective surgical therapy for select Dystonia patients who are refractory to medications or who have generalized symptoms (e.g. patients with Early-Onset Primary Dystonia(DYT1) mutations and other dystonia subtypes). DBS patients typically experience significant improvement in disabling symptoms; however, detailed programming is always required, and stimulation-induced side effects commonly emerge. Clinicians may empirically vary voltage, pulse width, frequency and also the active contacts on the DBS lead to achieve observed optimal benefits.

The majority of DBS patients undergo repeat surgeries to replace the implantable pulse generator (IPG) every 2.5 to 5 years. It has been demonstrated that, in dystonia patients, that higher settings are required for adequate symptomatic control, and that neurostimulators have a considerably shorter life when compared to neurostimulators from patients with essential tremor or Parkinson's disease. Additionally, several smaller studies have suggested that alternative pulse stimulation properties and pulse shape modifications can lower IPG battery consumption.

Newer patterns of stimulation (regularity of pulses and shapes of pulses) have not been widely tested in clinical practice, and are not part of the current FDA device labeling. Novel patterns of stimulation do however, have the potential to improve symptoms, reduce side effects, and to preserve the neurostimulator life.

The current research proposal will prospectively study biphasic pulse stimulation paradigms and its effects on dystonic symptoms. The investigators aim to demonstrate that we can tailor DBS settings to address dystonia symptoms, improve the safety profile, characterize distinct clinical advantages, and carefully document the safety and neurostimulator battery consumption profile for biphasic stimulation.

DETAILED DESCRIPTION:
In this research study, different stimulation patterns on the DBS device will be tried for effectiveness against current symptoms. There will be two different stimulation patterns that will be performed and can occur at different clinic dates. Each of the stimulation patterns will have times varying between 2-3 hours per stage. One part of the study will deliver stimulation in a continuous manner, while the other part of the study will deliver stimulation based upon responses obtained from changes in brain wave patterns. These procedures can be performed while in the clinic for regular programming visits or at different visits. The current DBS setting will be recorded and at the end of the session the setting will be reset to back to the previous settings. The participant will have the option of participating in both or just one part.

During the visit, the participant will be analyzed for tremor and slowness by using the Trigno wireless Electromyography (EMG) and the Kinesia system. The system includes a unit composed of two modules: a wrist module, which is the size of an I-Pod and will be attached to the wrist over a comfortable wristband, and a sensor module, which will be placed over the index finger.

The entire visit will be videotaped and UDRS (Unified Dystonia Disease Rating Scale) and BFMDRS (Burke-Fahn-Marsden Dystonia Rating Scale) scores will be evaluated by two scorers. Pre-DBS "off" and "on" scores will also be taken.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary generalized dystonia or cervical dystonia
* Bilaterally implanted globus pallidus interus(GPi) DBS.
* Minimum of 6 months of chronic stimulation
* Greater than 60 days on stable DBS settings

Exclusion Criteria:

* Does not have DBS for dystonia or cervical dystonia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a preliminary pilot investigation that will utilize a within subjects study design and will screen 10 generalized dystonia and screen 10 cervical dystonia patients.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-07; Primary Completion 2016-01 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Blinded Unified Dystonia Rating Scale (UDRS) | Day 1
  Neurologist use the UDRS to determine the severity and duration of dystonia on 14 body areas. Each body region is assessed and scores range from 0 (no dystonia) to 4 (extreme dystonia). The maximum UDRS score is 112 and includes severity and duration factors.
Burke-Fahn-Marsden Dystonia Rating Scale (BFMDRS) | Day 1
  Neurologist use the BFMDRS to rate the severity of dystonia in 9 regions of the body. Provoking and severity factors are ranked from 0 (no dystonia) to 4 (extreme dystonia) for each body region and then adjusted scores are summed to give an overall score from 0 to 120.

SECONDARY OUTCOMES:
Tremor accelerometer to measure motor dysfunction | Day 1
  Tremor accelerometer for the patients with a component of dystonic tremor (device taped or attached to the wrist by an elastic band to record how fast the tremor).
Kinesia accelerometer to measure motor dysfunction | Day 1
  Kinesia accelerometer for the patients with a mobile component of dystonia (device attached to the arms and legs (by an elastic band or tape) to record movements).
Battery Consumption compared between pre and post settings | Day 2
  Battery consumption will be calculated and compared between the NEW settings and patients' baseline settings. The Medtronic battery estimator helpline will be used to calculate battery life, as well as the University of Florida calculator.
GaitRite walking assessment. | Day 1
  The GaitRite is an automated floor that when you walk on the floor it records your gait pattern.

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Almeida, MD, Principal Investigator — University of Florida Center for Movement Disorders and Neurorestoration
Locations (1):
- Center for Movement Disorders and Neurorestoration, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Fakhar K, Hastings E, Butson CR, Foote KD, Zeilman P, Okun MS. Management of deep brain stimulator battery failure: battery estimators, charge density, and importance of clinical symptoms. PLoS One. 2013;8(3):e58665. doi: 10.1371/journal.pone.0058665. Epub 2013 Mar 11. PMID 23536810
- [Background] Rawal PV, Almeida L, Smelser LB, Huang H, Guthrie BL, Walker HC. Shorter pulse generator longevity and more frequent stimulator adjustments with pallidal DBS for dystonia versus other movement disorders. Brain Stimul. 2014 May-Jun;7(3):345-9. doi: 10.1016/j.brs.2014.01.008. Epub 2014 Jan 18. PMID 24548586
- [Background] Foutz TJ, McIntyre CC. Evaluation of novel stimulus waveforms for deep brain stimulation. J Neural Eng. 2010 Dec;7(6):066008. doi: 10.1088/1741-2560/7/6/066008. Epub 2010 Nov 17. PMID 21084732
- [Background] Hofmann L, Ebert M, Tass PA, Hauptmann C. Modified pulse shapes for effective neural stimulation. Front Neuroeng. 2011 Sep 28;4:9. doi: 10.3389/fneng.2011.00009. eCollection 2011. PMID 22007167
- [Background] Brocker DT, Grill WM. Principles of electrical stimulation of neural tissue. Handb Clin Neurol. 2013;116:3-18. doi: 10.1016/B978-0-444-53497-2.00001-2. PMID 24112880
- [Background] Birdno MJ, Kuncel AM, Dorval AD, Turner DA, Gross RE, Grill WM. Stimulus features underlying reduced tremor suppression with temporally patterned deep brain stimulation. J Neurophysiol. 2012 Jan;107(1):364-83. doi: 10.1152/jn.00906.2010. Epub 2011 Oct 12. PMID 21994263
- [Background] Swan BD, Grill WM, Turner DA. Investigation of deep brain stimulation mechanisms during implantable pulse generator replacement surgery. Neuromodulation. 2014 Jul;17(5):419-24; discussion 424. doi: 10.1111/ner.12123. Epub 2013 Oct 7. PMID 24118257
- [Background] Beuter A, Lefaucheur JP, Modolo J. Closed-loop cortical neuromodulation in Parkinson's disease: An alternative to deep brain stimulation? Clin Neurophysiol. 2014 May;125(5):874-85. doi: 10.1016/j.clinph.2014.01.006. Epub 2014 Jan 18. PMID 24555921
- [Background] Okun MS, Foote KD, Wu SS, Ward HE, Bowers D, Rodriguez RL, Malaty IA, Goodman WK, Gilbert DM, Walker HC, Mink JW, Merritt S, Morishita T, Sanchez JC. A trial of scheduled deep brain stimulation for Tourette syndrome: moving away from continuous deep brain stimulation paradigms. JAMA Neurol. 2013 Jan;70(1):85-94. doi: 10.1001/jamaneurol.2013.580. PMID 23044532
- See also: University of Florida Center for Movement Disorders & Neurorestoration — http://movementdisorders.ufhealth.org/